CLINICAL TRIAL: NCT00863564
Title: Acute Effects of Dietary Proteins on Postprandial Lipemia, Incretin Responses and Subclinical Inflammation in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Obesity Research Centre (Other); Nordic Centre of Excellence (Other)
Responsible Party: Kjeld Hermansen, Professor, Chief Physician, MD, Dr.Med.Sci, Department of Endocrinology And Metabolism, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CERN-PPL-JHJ-5a
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Obesity; Postprandial Lipemia; Atherosclerosis; Inflammation; Postprandial Incretins
Keywords: Postprandial Period; Postprandial Lipaemia; Incretins; Subclinical Inflammation; Obesity; Atherosclerosis; Triglyceride; Lipoproteins; Postprandial inflammation
MeSH Terms: conditions — Obesity; Atherosclerosis; Inflammation | interventions — CVD protocol; Glutens

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Whey Isolate (Active Comparator)
  Interventions: Dietary Supplement: Whey Isolate
- Caseine (Active Comparator)
  Interventions: Dietary Supplement: Caseine
- Cod (Active Comparator)
  Interventions: Dietary Supplement: Cod
- Gluten (Active Comparator)
  Interventions: Dietary Supplement: Gluten

INTERVENTIONS:
Dietary Supplement: Caseine
  Arms: Caseine
Dietary Supplement: Cod
  Arms: Cod
Dietary Supplement: Gluten
  Arms: Gluten
Dietary Supplement: Whey Isolate
  Arms: Whey Isolate

SUMMARY:
The purpose of this study is to determine the effects of dietary protein on blood lipids and gut hormones after a fat-rich meal.

Hypothesis: Certain dietary proteins reduce the amount of fat circulating in the blood stream following a fat rich meal. The effect is dependant of both the quality and the quantity of protein ingested.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2 & < 45 kg/m2

Exclusion Criteria:

* Diabetes
* Lipid lowering drugs
* Liver-, Kidney- and/or Heart Disease
* Serious Hypertension (160/110)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Triglyceride | 0h- 2h- 4h- 6h- 8h postprandial

SECONDARY OUTCOMES:
Incretins | 0h -1h -2h -4h -6h -8h Postprandial
Inflammatory markers | 0h- 1h- 2h- 4h- 6h- 8h postprandial

CONTACTS AND LOCATIONS:
Overall Officials: K Hermansen, Professor, MD, Principal Investigator — Department of Endocrinology and Metabolism, Aarhus University Hospital
Locations (1):
- Department of Clinical Nutrion, Aarhus, Denmark

REFERENCES:
- [Derived] Holmer-Jensen J, Karhu T, Mortensen LS, Pedersen SB, Herzig KH, Hermansen K. Differential effects of dietary protein sources on postprandial low-grade inflammation after a single high fat meal in obese non-diabetic subjects. Nutr J. 2011 Oct 19;10:115. doi: 10.1186/1475-2891-10-115. PMID 22011432